CLINICAL TRIAL: NCT05887960
Title: Impact of Neutrophil Lymphocyte and Monocyte Lymphocyte Ratio on Chronic Kidney Disease Patients Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdel rahman Hassan Mohamed, Impact of neutrophil lymphocyte and monocyte lymphocyte ratio on chronic kidney disease patients outcome, Assiut University
Other Study IDs: CKD patients
Record Dates: First submitted 2023-04-25; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Hemodialysis Complication
MeSH Terms: interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: healthy persons to see normal ratio of of neutrophil lymphocyte and monocyte lymphocyte
  Interventions: Other: CBC and flow cytometry test for monocyte
- 2: CKD patients stage (4-5) not on dialysis to see impact of (NLR) and (MLR) as regard inflamation and cardiovascular complications
  Interventions: Other: CBC and flow cytometry test for monocyte
- 3: patients ESRD on maintenance hemodialysis compared with CKD pre dialysis patents and see if hemodialysis is better for removal toxic granules and inflamatory markers caused by CKD
  Interventions: Other: CBC and flow cytometry test for monocyte

INTERVENTIONS:
Other: CBC and flow cytometry test for monocyte — all groups assigned Cbc with leukocyte differential and flow cytometry for monocyte population

SUMMARY:
The aim of this study is to establish NLR, MLR as a good predictors for outcome of CKD including hemodialysis and CKD stage (4-5) patients as regard inflammation, malnutrition and anemia on cardiovascular complication.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a global public health problem. With the decline in renal function, patients with end-stage kidney disease (ESKD) can choose hemodialysis (HD), peritoneal dialysis (PD) or kidney transplantation as renal replacement therapy to improve their quality of life. Globally, HD is still the most important renal replacement therapy.

With the continuous development and optimization of dialysis technology, the survival time of maintenance hemodialysis (MHD) patients is gradually prolonged. However, even in developed countries, the mortality rate of MHD patients remains high. According to data from the United States Renal Data System (USRDS) in 2019, the MHD mortality rate in 2017 was 167 per 1,000 patient-years.

Studies have shown that 30-50% of MHD patients have chronic inflammation state. Persistent inflammation can lead to a variety of complications, especially cardiovascular disease, malnutrition and anemia, thereby increasing the mortality of MHD patients.

Although less than 5% of MHD patients die directly from inflammation, inflammation can interact with a variety of risk factors and has an important impact on the prognosis of MHD patients. Studies have found that inflammation is closely related to high-risk factors of death such as myocardial hypertrophy, ventricular dysfunction, atherosclerosis, protein energy consumption, anemia and renal bone disease .

Therefore, the development of inflammation-related indicators has important clinical value for judging the prognosis of MHD patients and guiding early intervention.

Disturbed functions of polymorphonuclear leukocytes [PMNLs] lead to an enhanced risk of bacterial infections and represent a main cause for the increased risk of morbidity and mortality among CKD patients.

After chemotactic movement to the source of infection, PMNLs take up the invading microorganisms by phagocytosis and kill them with toxic oxygen radicals formed during the oxidative burst and proteolytic enzymes intracellularly released from granula.

Disturbances of any of those crucial PMNL functions increase the risk for bacterial infections. The proneness of CKD patients to infections resulting from decreased phagocytosis is caused by factors such as uremic toxins, iron overload, anemia of renal disease, and dialyzer bioincompatibility.

Neutrophils from HD patients show significantly elevated levels of reactive oxygen species (ROS) production, degranulation, and basal neutrophil extracellular trap (NET) formation, indicating spontaneous activation.

Furthermore, similar to PMNLs from patients with acute infections. Monocytes are bone marrow derived cells that circulate in the blood for 1-3 days before differentiating into tissue macrophages or dendritic cells. In a review in this special issue, Girndt et al.

focuses on the differences of uremic monocytes in the expression of surface molecules, the production of cytokines and mediators, and in their function as compared to monocytes of healthy persons.

Based on their CD14/CD16 expression profile, three distinct populations of monocytes can be distinguished: Mo1 ("classical monocytes" expressing CD14 only), Mo2 ("intermediate monocytes", CD14++/CD16+), and Mo3 ("non-classical monocytes", CD14+/CD16++). The Mo2 population has pronounced pro-inflammatory properties. Their proportion is an important predictor of mortality risk in HD patients [35].

The contribution of monocytes to the dysregulated immune response in uremia can be based on altered features of the individual cells or on a change in the relative numbers of the three different populations. Monocytes play an important role in both innate immunity and antigen presentation for specific cellular immune defense.

In patients with chronic renal failure as well as those treated with maintenance hemodialysis, these cells are largely dysregulated.

Monocytes and macrophages strongly contribute to the pathogenesis of atherosclerosis. These cells invade the vessel wall at sites of endothelial lesions and participate in the formation of foam cells, the deposition of lipids in the intima, and the growth of the atheromatous plaque. Macrophages within vascular plaques express inflammatory markers .

These observations prompted the study of a relationship between the activation of circulating monocytes in the blood of dialysis patients and their risk of atherosclerotic vascular disease. Investigators found many hints that such relation exists. Studies in dialysis patients described correlations between monocyte expression of IL-1 and IL-1RA and cardiovascular events.

The relative frequency of CD14++/16+ Mo2 cells relates to this morbidity in different cohorts with CKD including HD, PD and CKD patients stages 1-5 [37,35,33].

A high expression of ACE on monocytes appears to be associated with cardiovascular disease in HD and PD patients.

In addition, the intensity of monocyte sequestration during a dialysis session as a surrogate for the activation level of this cell type is predictive for cardiovascular events as well.

Since many of the morphological and functional alterations of monocytes are found in both CKD 3-5 and dialysis patients, uremic toxicity may be one of the important causal factors.

However, hemodialysis accentuates some of the monocyte abnormalities. This might be the consequence of inflammatory activation through blood-membrane interactions, and biocompatibility issues may play a role.

Further, dialysis can clear several but not all retention solutes from the blood of uremic patients. It is thus reasonable to test different dialysis modalities (HDF, high cut-off dialysis) if they influence monocyte dysfunction. All these aspects have been addressed in clinical or experimental studies.

Recent studies have found that the ratios of different blood cell components are new inflammatory markers, which have good predictive value in the outcome of CKD, cardiovascular disease, rheumatic disease, etc., including neutrophil-to-lymphocyte ratio (NLR) , monocyte-to-lymphocyte ratio (MLR) , Previous studies have inconsistent conclusions about the predictive value of NLR and MLR on mortality of HD patients. Xiang et al. suggested that higher MLR was a strong and independent predictor of all-cause and cardiovascular mortality and overwhelmed NLR among HD patients .

This study hypothesized that the combination of NLR and MLR could form a new indicator for predicting the mortality of HD patients. Therefore, the study incorporated NLR and MLR into an inflammation scoring system and investigated the value of inflammation score in predicting all-cause and cardiovascular mortality in HD patients.

Besides neutrophil and lymphocytes, monocytes play a key role in inflammation and are well known as a central factor in pathogenesis of atherosclerosis. Patients with ESRD exhibit a general expansion of circulating monocytes with increased basal production of cytokines and reactive oxygen species (ROS), which contribute to the prevailing oxidative stress and systemic inflammation in this population. On the other hand, this kind of spontaneous activation is accompanied by decreased phagocytic capacity of monocytes and impaired antigen presentation capacity, thus leading to defective functions of T and B cells; the impaired expression of co-stimulatory molecules also contributes to this phenomenon. Findings from epidemiological studies indicate that elevated monocyte counts are independently related to all-cause and cardiovascular mortality in HD patients.

ELIGIBILITY:
Inclusion Criteria:

* - Hemodialysis patients > 18 years
* < 60 years old
* CKD stage (4-5) not on dialysis

Exclusion Criteria:

* o Recent acute coronary or cerebrovascular accident

  * Autoimmune diseases
  * Hematological diseases
  * Liver cirrhosis
  * Active or pre-active infection
  * Malignancy
  * Medications as Aspirin, NSAI, immunosuppressive steroid.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy persons as control group patients with chronic kidney disease (CKD) stage 4-5 (not on dialysis) patients ESRD on maintenance hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Impact of neutrophil lymphocyte and monocyte lymphocyte ratio on chronic kidney disease patients outcome | baseline
  Neutrophil to lymphocyte ratio and monocyte to lymphocyte ratio in addition to subtypes of monocytes will be measured in healthy persons, CKD patients stage (4-5) and in chronic hemodialysis patients and use it as inflamamtory markers as well as it's a good predictors for cardiovascular complications and what's the impact of it's ratio degree on CKD patients outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf AN el shazly, profeassor, Principal Investigator — Assiut University

REFERENCES:
- [Background] Kim JK, Hong CW, Park MJ, Song YR, Kim HJ, Kim SG. Increased Neutrophil Extracellular Trap Formation in Uremia Is Associated with Chronic Inflammation and Prevalent Coronary Artery Disease. J Immunol Res. 2017;2017:8415179. doi: 10.1155/2017/8415179. Epub 2017 Mar 27. PMID 28523279
- [Background] Girndt M, Trojanowicz B, Ulrich C. Monocytes in Uremia. Toxins (Basel). 2020 May 21;12(5):340. doi: 10.3390/toxins12050340. PMID 32455723
- [Result] Ramirez R, Carracedo J, Merino A, Soriano S, Ojeda R, Alvarez-Lara MA, Martin-Malo A, Aljama P. CD14+CD16+ monocytes from chronic kidney disease patients exhibit increased adhesion ability to endothelial cells. Contrib Nephrol. 2011;171:57-61. doi: 10.1159/000327134. Epub 2011 May 23. PMID 21625090
- [Result] Chapter 1: Definition and classification of CKD. Kidney Int Suppl (2011). 2013 Jan;3(1):19-62. doi: 10.1038/kisup.2012.64. No abstract available. PMID 25018975
- [Result] Kato S, Chmielewski M, Honda H, Pecoits-Filho R, Matsuo S, Yuzawa Y, Tranaeus A, Stenvinkel P, Lindholm B. Aspects of immune dysfunction in end-stage renal disease. Clin J Am Soc Nephrol. 2008 Sep;3(5):1526-33. doi: 10.2215/CJN.00950208. Epub 2008 Aug 13. PMID 18701615
- [Result] Sarnak MJ, Jaber BL. Mortality caused by sepsis in patients with end-stage renal disease compared with the general population. Kidney Int. 2000 Oct;58(4):1758-64. doi: 10.1111/j.1523-1755.2000.00337.x. PMID 11012910
- [Result] Mansur A, Mulwande E, Steinau M, Bergmann I, Popov AF, Ghadimi M, Beissbarth T, Bauer M, Hinz J. Chronic kidney disease is associated with a higher 90-day mortality than other chronic medical conditions in patients with sepsis. Sci Rep. 2015 May 21;5:10539. doi: 10.1038/srep10539. PMID 25995131
- [Result] James MT, Laupland KB, Tonelli M, Manns BJ, Culleton BF, Hemmelgarn BR; Alberta Kidney Disease Network. Risk of bloodstream infection in patients with chronic kidney disease not treated with dialysis. Arch Intern Med. 2008 Nov 24;168(21):2333-9. doi: 10.1001/archinte.168.21.2333. PMID 19029498
- [Result] Haag-Weber M, Horl WH. Dysfunction of polymorphonuclear leukocytes in uremia. Semin Nephrol. 1996 May;16(3):192-201. PMID 8734462
- See also: He, T.; Xiong, J.; Huang, Y.; Zheng, C.; Liu, Y.; Bi, X.; Liu, C.; Han, W.; Yang, K.; Xiao, T.; et al. Klotho restrain RIG-1/NF-κB signaling activation and monocyte inflammatory factor release under uremic condition. Life Sci — http://scholar.google.com/scholar_lookup?title=Klotho+restrain+RIG-1/NF-%CE%BAB+signaling+activation+and+monocyte+inflammatory+factor+release+under+uremic+condition&author=He,+T.&author=Xiong,+J.&author=Huang,+Y.&author=Zheng,+C.&author=Liu,+Y.&author=Bi,+X.&author=Liu,+C.&author=Han,+W.&author=Yang,+K.&author=Xiao,+T.&publication_year=2019&journal=Life+Sci.&volume=231&pages=116570&doi=10.1016/j.lfs.2019.116570